CLINICAL TRIAL: NCT04853641
Title: The Impact of Advanced Age and High BMI on Short-term Outcomes in Live-donor Liver Transplant Recipients
Brief Title: Impact of Age and BMI on Liver Transplant Outcomes
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ibtesam Hilmi, Professor, University of Pittsburgh
Other Study IDs: STUDY20070432
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Liver Transplant; Complications; Perioperative/Postoperative Complications
Keywords: Age Related Outcomes; BMI related outcomes; Liver Transplantation
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Living Donor Liver Transplant Recipient: Patients who have received a living donor liver transplant.
  Interventions: Procedure: Living Donor
- Deceased Donor Liver Transplant Recipient: Patients who have received either a Deceased by Circulatory Death or Deceased by Brain Death Liver Transplant
  Interventions: Procedure: Cadaveric

INTERVENTIONS:
Procedure: Cadaveric — Cadaveric Organ Transplant
  Groups: Deceased Donor Liver Transplant Recipient
Procedure: Living Donor — Living Donor Organ Transplant
  Groups: Living Donor Liver Transplant Recipient

SUMMARY:
Prospectively enrolled retrospective chart review and Liver Transplant database review to determine the modifiable and nonmodifiable risk factors specifically relating to Living Donor Liver Transplants. To observe the impact of age and BMI on graft outcomes and whether they impact the intraoperative management, post-operative length of stay, and complications.

DETAILED DESCRIPTION:
There has been a great deal of research into the characteristics of the donor for organ transplant, with older donors and those with more comorbidities having worse function once the organ is implanted. There has not been a great deal of research in the United States about the recipient's characteristic including age and BMI and the effects on donor organ function. With increasingly expanded criteria for organ recipients especially in the field of living donor organs the investigators plan to show the impact of older age and increased BMI on newly transplanted organs.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a liver transplant at UPMC- Montefiore Hospital Age> 18

Exclusion Criteria:

* Excludes Children (<18 years old) as they do not receive their operation under the same protocols Lost to follow-up prior to 1 year Participation in alternate research protocol that significantly altered the care they received in the perioperative period that may make their inclusion skew results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage liver disease, cirrhosis, or cancer requiring a liver transplant.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Graft Function 30 day | 30 day
  How well does the organ function
Mortality | 1 year
  Mortality at 1 year
Graft Survival 1 year | 1 year
  Survival of Organ at 1 year

SECONDARY OUTCOMES:
Perioperative Complications | 30 day
  Any complications in the perioperative period
Length of Stay- Total and ICU | Up to 6 months
  How long after surgery before patient is discharged from ICU and from Hospital
Duration of Intubation/Ventilation | Up to 6 months
  Time from Surgery End to Extubation or no longer requiring ventilatory support
Postoperative Complications | Up to 6 months
  Complications in the postoperative period- Renal, Infectious Disease, Pulmonary, Cardiac, Transplant related, Reintubation, Reoperation
Blood Transfusion | Up to 2 days
  Amount of blood transfusion required intraoperatively
Vasoactive Medication | Up to 2 days
  Amount and Type of Vasoactive Medication used at procedure end

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Montefiore, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No current plans